CLINICAL TRIAL: NCT05620719
Title: Project MARCH: Multisite Advancement of Research on Chronic Posttraumatic Headache
Brief Title: Multisite Advancement of Research on Chronic Posttraumatic Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); C.R.Darnall Army Medical Center (U.S. Federal Agency); Desmond Doss Health Clinic, Schofield Barracks (Unknown); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); South Texas Veterans Health Care System (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); Harvard University (Other); University of California, Los Angeles (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Donald McGeary, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20220592H
Record Dates: First submitted 2022-11-01; First posted 2022-11-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Headache
Keywords: Cognitive Behavioral Therapy; Telehealth; Veterans; Military Service Members; Chronic Pain; Headaches
MeSH Terms: conditions — Post-Traumatic Headache; Chronic Pain; Headache | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Independent evaluators will complete posttreatment and follow-up assessments with each participant. They will instruct participants not to share which treatment group they were assigned. The Principle Investigator will remain blind to treatment randomization outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinic-based Cognitive Behavioral Therapy (CCBT) (Active Comparator): CCBT provides CBT for posttraumatic headache through 8 face-to-face, in-clinic sessions.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Posttraumatic Headache
- Telemedicine-based Cognitive Behavioral Therapy (TCBT) (Active Comparator): TCBT provides 8-sessions of CBT for posttraumatic headache using telemedicine technology rather than attending in-office sessions. Additionally, TCBT includes instructions for each session specific to the mechanics of a telehealth encounter (e.g., asking participant for name, location, and accessible phone number for location in case of technical failure or crisis). All TCBT participants must be enrolled at the MTF or VA from which they were recruited, and the treatment facility will be notified that they are receiving TCBT in case a crisis arises and needs to be managed by the site.
  Interventions: Other: Telemedicine-based Cognitive Behavioral Therapy (TCBT)
- Treatment As Usual (Active Comparator): Participants will continue to engage in clinical care as usual for 8 weeks. Research staff will call the TAU participants weekly to assess for adverse events. Research staff at each site will be trained on standardized assessment of usual care activities using forms adapted from our single-site trial.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Posttraumatic Headache — CBT for Posttraumatic Headaches consists of 8 sessions of cognitive behavioral therapy that focus on (1) discussions and exercises that increase awareness of what may be related to headaches, (2) relaxation techniques to manage physiological stress, and (3) problem-solving techniques to manage common stressors. Sessions are delivered weekly and can last between 45 to 75 minutes based on clinical content and patient response to the material.
  Other Names: CCBT
  Arms: Clinic-based Cognitive Behavioral Therapy (CCBT)
Other: Treatment as Usual — Participants will continue to engage in medical care as usual for 8 weeks.
  Other Names: TAU or TPU
  Arms: Treatment As Usual
Other: Telemedicine-based Cognitive Behavioral Therapy (TCBT) — Participants assigned to TCBT will receive 8 sessions of cognitive behavioral therapy using telemedicine rather than face-to face office visits.
  Arms: Telemedicine-based Cognitive Behavioral Therapy (TCBT)

SUMMARY:
Posttraumatic headache (PTH) is a common and highly disabling consequence of traumatic brain injury (TBI) in U.S. military service members and veterans. Cognitive Behavioral Therapy for PTH has been shown to significantly improve disability outcomes in veterans with persistent PTH when delivered in-person. Telemedicine platforms can dramatically increase access to evidence-based care. However, whether CBT for PTH retains its effectiveness when delivered through a telemedicine platform has yet to be established. The purpose of this 3-arm randomized clinical trial is to compare Clinic-based Cognitive-Behavioral Therapy (CCBT) to Telemedicine-based Cognitive Behavioral Therapy (TCBT) and to treatment as usual (TAU) in 525 service members and veterans with chronic posttraumatic headaches (PTH) at 4 VA medical centers* and 3 military treatment facilities across the U.S. Participants will be assessed for headache-related disability, headache experience, and psychiatric comorbidities across multiple time points.

*VA Palo Alto Health Care System is temporarily randomizing into TAU and TCBT only.

DETAILED DESCRIPTION:
Posttraumatic headache (PTH) is noticeably more common among military service members and veterans than among civilians, with an estimated 80-90% of veterans with TBI reporting new or exacerbated headaches. Unlike civilian PTH, military and veteran PTH is likely to become chronic and recalcitrant to most front-line interventions for primary headache (e.g., migraine, tension-type). Service members and veterans with PTH report significantly decreased productivity in work and home activities and high rates of military discharge and work absenteeism. Pharmacological treatments for chronic PTH have proven problematic (i.e., unwanted side effects; worsening of symptoms long term). However, prior to 2019, guidance for non-pharmacological treatment approaches for PTH was unclear. In 2019, the investigators completed a single-site randomized clinical trial comparing Clinic-based CBT for PTH to Treatment at Usual in 193 veterans with PTH. The study found that Clinic-based CBT for PTH led to a significant improvement in headache-related disability (as measured by the 6-Item Headache Impact Test; HIT-6) at follow-up. In contrast, headache disability scores for participants in the Treatment as Usual condition remained unchanged.

COVID-19 pandemic led to widespread recognition of the need for distance-technology platforms to add meaningful infrastructure for extended service delivery without the limitations of in-office care. Telehealth-based care can decrease the cost and increase the convenience of treatment leading some to suggest that telehealth may eventually become a first option for treating patients. Given the potential impact of CBT for PTH to improve the functioning of service members and veterans with PTH following TBI, it is important to determine whether the results of the single-site trial can be replicated across diverse geographic regions and whether CBT for PTH retains its efficacy in improving headache-related disability when delivered through telemedicine platforms.

The study has four aims.

Aim 1: Determine the efficacy of Clinic-based Cognitive-Behavioral Therapy (CCBT; using our manualized intervention) and Telemedicine-Based Cognitive Behavioral Therapy (TCBT; using our manualized intervention) for posttraumatic headache (PTH) compared to treatment as usual (TAU) across seven geographically-dispersed treatment sites.

Hypothesis 1A: There will be significantly greater improvement in PTH disability (measured by the Headache Impact Test-6; HIT-6) at 3-month follow-up among service members and veterans in CCBT compared to TAU.

Hypothesis 1B: There will be significantly greater improvement in PTH disability (measured by the HIT-6) at 3-month follow-up for service members/veterans who participate in TCBT compared to TAU.

Aim 2: Establish the non-inferiority of TCBT to CCBT in the treatment of PTH-related disability. This second aim will be pursued if either CCBT or TCBT is superior to TAU in Aim 1.

Hypothesis 2: TCBT will be non-inferior to CCBT on headache-related disability (measured by the HIT-6) at 3-month follow-up.

Aim 3: Assess contribution of heterogeneity treatment effects on PTH treatment outcome. A patient-level model to assess heterogeneity treatment effect (HTE) based on site, system, and patient-level factors including all participants across sites will be run and the degree of benefit conditional on the model predictors using procedures from the Predictive Approaches to Treatment Effect Heterogeneity statement (PATH) will be assessed.

Hypothesis 3: A prognostic model consisting of baseline predictors will adequately predict disability risk with good precision and calibration. Individuals predicted to be at high risk of disability will exhibit differential treatment response, with less expected benefit than individuals with less risk.

Aim 4: Solicit participant perspectives on their treatment experience and identify patient-centered treatment targets that might better reflect their response to treatment.

Hypothesis 4A: Patients will identify measurable treatment targets across multiple domains.

Hypothesis 4B: Patients will provide treatment insights that might better reflect their response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any veteran or active duty service member (DEERS-eligible; age 18 to 70 years) with mild or moderate TBI whose headache began or exacerbated within 3 months of a head or neck injury.
* Headache meets ICHD-3 A5.2 criterion for delayed-onset persistent headache attributable to mild or moderate TBI and PTH is ongoing at enrollment (most recent headache within the past 2 weeks).
* At least moderate to severe headache-related disability based on a HIT-6 score greater than 50.
* Participant is stable on headache medication at baseline assessment (i.e., no changes in medication prescriptions in the past 4 weeks or study physician clinical judgement confirms stability; this includes botulinum toxin injections and devices like Cefaly).
* Participant has a phone where they can receive reminders and complete the on-line Headache Diaries.
* Participant speaks and reads/understands English well enough to fully participate in the intervention and to reliably complete assessment measures.

Exclusion Criteria:

* Participant reports a significant change in headache symptoms within 4 weeks of screening or has another secondary headache that may account for symptoms.
* Participant has medication overuse headache based on Structured Diagnostic Headache Interview-Revised (Brief Version; SDIH-R) and clinical judgment.
* Participant has a psychiatric problem that warrants immediate treatment as indicated in the electronic health record, flagged study during testing, or confirmed by a clinician through screening or review of clinical notes.
* Participant demonstrates significant cognitive impairment that could impact treatment adherence/benefit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Headache Impact Test (HIT-6) | Baseline to 3-month follow-up
  Headache-disability as measured by the Headache Impact Test. The HIT-6 is a 6-item measure of headache-disability. The measure uses a 5-point Likert scale to rate the frequency that the respondent experiences headache-relate disability across six domains of functioning. Total scores range from 36 to 78 with higher scores representing a higher level of headache-relate disability.

SECONDARY OUTCOMES:
Change in Standardized Headache Diary | Baseline to 3-month follow-up
  Headache frequency, duration and intensity will be assessed using a smartphone-based daily headache self-monitoring diary developed by the HCoE. During treatment, participants will record their headache intensity twice daily, using a 0 to 10 scale, to assess: (a) days per week with a headache (ranging from 0 to 7); (b) weekly headache frequency (range from 0 to 10); (c) headache duration (>= 0 hours); and (d) average peak headache intensity (range from 0 to 10).
Change in Patient Health Questionnaire-9 | Baseline to 3-month follow-up
  Total score on the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is 9-item, self-report screener for current depressive symptoms. Each item is rated on a frequency scale ranging from 0 (Not at all) to 3 (Nearly Every day). The measure provides a total severity score that ranges from 0 to 27, with higher scores representing more severe depressive symptoms.
Change in Generalized Anxiety Disorder Screener-7 | Baseline to 3-month follow-up
  Total score on the Generalized Anxiety Disorder Screener (GAD-7): The GAD-7 is 7-item, self-report screener for current anxiety symptoms. Each item is rated on a frequency scale ranging from 0 (Not at all) to 3 (Nearly Every day). The measure provides a total severity score that ranges from 0 to 21, with higher scores representing more severe anxiety symptoms.
Change in PTSD Checklist-5 | Baseline to 3-month follow-up
  Scale measurements by the PTSD CheckList-5 (PCL-5). The PCL-5 is a 20-item, self-report measure of PTSD symptoms experienced in the past month. Each item is rated on a severity scale ranging from 0 (Not at all) to 4 (Extremely). The measure provides a total severity score that ranges from 0 to 80, with higher scores representing more PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Donald D McGeary, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (8):
- United States (8):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Tripler Army Medical Center (Desmond Doss Health Clinic, Schofield Barracks), Honolulu, Hawaii
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - Carl R. Darnall Army Medical Center (Fort Cavazos), Killeen, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arcaya MC, Lowe SR, Asad AL, Subramanian SV, Waters MC, Rhodes J. Association of posttraumatic stress disorder symptoms with migraine and headache after a natural disaster. Health Psychol. 2017 May;36(5):411-418. doi: 10.1037/hea0000433. Epub 2016 Dec 8. PMID 27929328
- [Background] Cameron IM, Crawford JR, Lawton K, Reid IC. Psychometric comparison of PHQ-9 and HADS for measuring depression severity in primary care. Br J Gen Pract. 2008 Jan;58(546):32-6. doi: 10.3399/bjgp08X263794. PMID 18186994
- [Background] Dave A, Ganesh A, Adil MM, Tsao JW. Practice Current: How do you diagnose and treat post-concussive headache? Neurol Clin Pract. 2019 Jun;9(3):263-270. doi: 10.1212/CPJ.0000000000000656. PMID 31341715
- [Background] Eckner JT, Seifert T, Pescovitz A, Zeiger M, Kutcher JS. Is Migraine Headache Associated With Concussion in Athletes? A Case-Control Study. Clin J Sport Med. 2017 May;27(3):266-270. doi: 10.1097/JSM.0000000000000346. PMID 27428679
- [Background] Holtkamp MD, Grimes J, Ling G. Concussion in the Military: an Evidence-Base Review of mTBI in US Military Personnel Focused on Posttraumatic Headache. Curr Pain Headache Rep. 2016 Jun;20(6):37. doi: 10.1007/s11916-016-0572-x. PMID 27084376
- [Background] Jaramillo CA, Eapen BC, McGeary CA, McGeary DD, Robinson J, Amuan M, Pugh MJ. A cohort study examining headaches among veterans of Iraq and Afghanistan wars: Associations with traumatic brain injury, PTSD, and depression. Headache. 2016 Mar;56(3):528-39. doi: 10.1111/head.12726. Epub 2015 Dec 21. PMID 26688427
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Lew HL, Lin PH, Fuh JL, Wang SJ, Clark DJ, Walker WC. Characteristics and treatment of headache after traumatic brain injury: a focused review. Am J Phys Med Rehabil. 2006 Jul;85(7):619-27. doi: 10.1097/01.phm.0000223235.09931.c0. PMID 16788394
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] McGeary DD, McGeary CA, Gatchel RJ. A comprehensive review of telehealth for pain management: where we are and the way ahead. Pain Pract. 2012 Sep;12(7):570-7. doi: 10.1111/j.1533-2500.2012.00534.x. Epub 2012 Feb 5. PMID 22303839
- [Background] McGeary DD, McGeary CA, Gatchel RJ, Allison S, Hersh A. Assessment of research quality of telehealth trials in pain management: a meta-analysis. Pain Pract. 2013 Jun;13(5):422-31. doi: 10.1111/j.1533-2500.2012.00601.x. Epub 2012 Sep 27. PMID 23017210
- [Background] McGeary DD, Penzien DB, Resick PA, McGeary CA, Jaramillo CA, Eapen BC, Young-McCaughan S, Nabity PS, Moring JC, Houle TT, Keane TM, Peterson AL. Study design for a randomized clinical trial of cognitive-behavioral therapy for posttraumatic headache. Contemp Clin Trials Commun. 2021 Jan 6;21:100699. doi: 10.1016/j.conctc.2021.100699. eCollection 2021 Mar. PMID 33490706
- [Background] Minen M, Jinich S, Vallespir Ellett G. Behavioral Therapies and Mind-Body Interventions for Posttraumatic Headache and Post-Concussive Symptoms: A Systematic Review. Headache. 2019 Feb;59(2):151-163. doi: 10.1111/head.13455. Epub 2018 Dec 1. PMID 30506568
- [Background] Roper LS, Nightingale P, Su Z, Mitchell JL, Belli A, Sinclair AJ. Disability from posttraumatic headache is compounded by coexisting posttraumatic stress disorder. J Pain Res. 2017 Aug 21;10:1991-1996. doi: 10.2147/JPR.S129808. eCollection 2017. PMID 28860853
- [Background] Schwedt TJ, Dodick DW, Hentz J, Trentman TL, Zimmerman RS. Occipital nerve stimulation for chronic headache--long-term safety and efficacy. Cephalalgia. 2007 Feb;27(2):153-7. doi: 10.1111/j.1468-2982.2007.01272.x. PMID 17257236
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Theeler BJ, Flynn FG, Erickson JC. Headaches after concussion in US soldiers returning from Iraq or Afghanistan. Headache. 2010 Sep;50(8):1262-72. doi: 10.1111/j.1526-4610.2010.01700.x. Epub 2010 Jun 10. PMID 20553333